CLINICAL TRIAL: NCT00532532
Title: AV650-018: A Two-Part (Double-Blind Followed by Open-Label), Placebo Controlled, Randomized Trial to Assess the Safety, Tolerability, and Preliminary Efficacy of AV650 (Tolperisone HCl) in Subjects With Spasticity Associated With Multiple Sclerosis
Brief Title: Safety and Preliminary Effectiveness of AV650 in Patients With Spasticity Associated With Multiple Sclerosis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Avigen (Industry)
Responsible Party: Glenn Morrison, Ph.D., Avigen, Inc.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AV650-018
Record Dates: First submitted 2007-09-18; First posted 2007-09-20 (Estimated); Last update posted 2008-11-04 (Estimated); Status verified 2008-11

CONDITIONS: Muscle Spasticity
Keywords: Multiple sclerosis
MeSH Terms: conditions — Muscle Spasticity; Multiple Sclerosis | interventions — Tolperisone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): AV650 low dose
  Interventions: Drug: tolperisone HCl
- 2 (Experimental): AV650 high dose
  Interventions: Drug: tolperisone HCl
- 3 (Experimental): Placebo
  Interventions: Drug: tolperisone HCl

INTERVENTIONS:
Drug: tolperisone HCl — Low dose AV650 three times a day orally for 5 weeks; followed by optional continuation on either low dose or high dose AV650, as tolerated, for 24 weeks
  Arms: 1
Drug: tolperisone HCl — High dose AV650 three times a day orally for 5 weeks; followed by optional continuation on either low dose or high dose AV650, as tolerated, for 24 weeks
  Arms: 2
Drug: tolperisone HCl — Placebo three times a day orally for 5 weeks; followed by optional continuation on either low dose or high dose AV650, as tolerated, for 24 weeks
  Arms: 3

SUMMARY:
A drug called AV650 (tolperisone HCl) will be given to patients who have spasticity associated with multiple sclerosis. This study has three purposes:

1. To determine whether AV650 is safe for patients with multiple sclerosis;
2. To gather some early evidence as to whether AV650 is effective in treating spasticity in patients with multiple sclerosis; and,
3. To assess what the body does with AV650 once it is ingested (Germany and Czech Republic sites only).

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects between 18 and 70 years of age (inclusive)
* Signed and dated informed consent
* Definite MS as per Poser or MacDonald Criteria (either relapsing remitting or secondary progressive course)
* Expanded Disability Status Score (EDSS) from 3.0 to 6.5 (inclusive) at Screening
* Stable MS for at least 30 days before screening
* Female of child bearing potential and male subjects whose partner is of child bearing potential who are willing to ensure that they or their partner use effective double-barrier contraception during the study and for 90 days thereafter
* If female, be neither pregnant nor nursing (Confirmation that the subject is not pregnant must be established by a negative serum hCG pregnancy test at baseline.)
* Significant spasticity in at least two muscle groups defined as a score of 2 or more on the Ashworth scale for each muscle group
* If a subject is on anti-spastic treatments, the dosage, frequency, and route of administration must be stable for at least 30 days before Screening
* If a subject is on MS treatments, the dosage, frequency, and route of administration must be stable for at least 30 days before Screening

Exclusion Criteria:

* Subjects who have participated in another research study within 90 days of Screening
* Significant changes in anti-spasticity medications (dosage, frequency, or route of administration) within 30 days of Screening
* Known hypersensitivity to tolperisone HCl, its components, or other lidocaine/lidocaine-like products
* Use of tolperisone HCl within 30 days of screening
* Significant changes in MS treatments (dosage, frequency, or route of administration) within 30 days of Screening
* Spasticity due to neurological disorders other than MS
* Any psychiatric disorder or cognitive impairment that precludes fully informed consent or safe participation in the study
* Subjects who have suffered an acute relapse of MS or who continue to suffer from an acute relapse of MS within 90 days of Baseline
* History of alcohol or substance abuse within one year of Screening
* Concurrent clinically significant immunologic, pulmonary, renal, hepatic, or endocrine disease and/or other unstable or major disease other than MS
* Clinically significant cardiovascular disorders, such as ischemic heart disease, arrhythmias, poorly controlled hypertension, or acute myocardial infarction
* QT prolongation greater than 480 msec or greater than 450 msec if accompanied by a partial bundle branch block, or other ECG abnormality in the judgment of the Investigator
* Diastolic blood pressure <50mmHg or >105mmHg; heart rate <50 beats per minute (bpm) or >110bpm, after 3 minutes in a sitting position; heart rate by ECG <50bpm or >110bpm
* History of epilepsy (except childhood febrile seizures)
* Current malignancy or history of malignancy that has not been in remission for more than five years, except basal cell skin carcinoma and cervical cancer (with treatment)
* Female subject who is pregnant, nursing, or planning pregnancy during the course of the study
* Scheduled elective surgery or other procedures requiring general anesthesia during the study
* Subject who is terminally ill in the judgment of the Investigator
* Subject who is inappropriate for placebo medication in the judgment of the Investigator
* Systemic corticosteroid therapy within 28 days of randomization, with the exception of inhaled medications for asthma
* Exacerbation of MS within 30 days of Baseline
* Regular levo-dopa therapy within 7 days of randomization
* Subjects taking antiarrhythmic medications
* Donation of blood during the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2007-09; Primary Completion 2008-09 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
To determine the long-term safety and tolerability of AV650 (tolperisone HCl) in subjects with spasticity associated with MS | 38 weeks

SECONDARY OUTCOMES:
To determine preliminary efficacy of AV650 as compared to placebo in subjects with spasticity associated with MS; and to determine the pharmacokinetic (PK) profile of AV650 at two dose levels | 38 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Glenn Morrison, MSc, PhD, Study Director — Avigen, Inc.
Locations (28):
- Czechia (4):
  - Annes University Hospital, Brno
  - University Hospital Hradec Kralove, Hradec Králové
  - University Hospital Plzen, Pilsen
  - University Hospital Motol, Prague
- Germany (9):
  - Facharzt fur Neurologie, Bad Saarow
  - Facharztin fur Neurologie und Psychiatrie, Berlin
  - Facharzt fur Neurologie und Psychiatrie, Berlin
  - Private practice, Berlin
  - Neurological practice, Bochum
  - Neurological practice, Cologne
  - Neuro-Consil GmbH, Düsseldorf
  - X-pert-med GmbH, Gräfelfing
  - Asklepios Klinik Nord-Heidberg, Hamburg
- Russia (5):
  - City Hospital #33, Nizhny Novgorod
  - Regional Clinical Hospital named Semashko, Nizhny Novgorod
  - Institute of Human Brain, Saint Petersburg
  - Leningrad Regional Clinical Hospital, Saint Petersburg
  - Nikolaevskaya Hospital, Complex Rehabilitation Department, Saint Petersburg
- Serbia (2):
  - Clinical Center of Serbia Institute of Neurology, Belgrade
  - Clinical Center Nis Clinic of Neurology, Niš
- Ukraine (8):
  - Ivano-Frankivsk Regional Clinical Hospital, Ivano-Frankivsk
  - Central Clinical Hospital Ukrzalinznytsi (Dept. Neur. No. 1), Kharkiv
  - Central Clinical Hospital Ukrzalinznytsi (Dept. Neur. No. 3), Kharkiv
  - Institute of Neurology, Psychiatry and Narcology of AMS of Ukraine, Kharkiv
  - Institute of Clinical Radiology of the Scientific Centre of Radiation Medicine of the AMS of Ukraine, Kyiv
  - Odesa Regional Psychoneurological Dispensary, Odesa
  - M.O.Semashko Republican Clinical Hospital, Simferopol
  - Uzhgorod Regional Centre of Neurosurgery and Neurology, Uzhhorod